CLINICAL TRIAL: NCT06769685
Title: TPO Combined With TPORA for Solid Tumors Effectiveness of cTit Above Degree II
Status: Enrolling by invitation | Type: Observational
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, jianfei Fu, chief physician, Jinhua Central Hospital
Other Study IDs: JinhuaCH
Record Dates: First submitted 2025-01-01; First posted 2025-01-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: CTIT-Chemotherapy Induced Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Information about patients will be collected prospectively in this study, which will collect information about all enrolled patients' two tumor treatment cycles and prothrombogenic drug therapy during them. The data to be collected will include the patient's baseline characteristics, the dose, frequency, and duration of each study drug, the name, dose, frequency, and duration of any combinations of study drugs, laboratory tests (e.g., blood counts) before, during, and after treatment with each study drug, and records of adverse events, including those related to the patients' baseline characteristics. and other relevant content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: For ctit patients with platelet counts ≥50×109/L and <75×109/L, they were randomized into groups A.
  Interventions: Drug: rhTPO; Drug: hypertrombopa
- Group B: For ctit patients with platelet counts <50×109/L, they were randomized into groups B.
  Interventions: Drug: rhTPO; Drug: hypertrombopa

INTERVENTIONS:
Drug: rhTPO — In group A, they were treated with rhTPO and hypertrombopa, and were medicated until their PLT was ≥75×109/L. In group B, they were treated with rhTPO and hypertrombopa, and were medicated until their PLT was ≥75×109/L.
Drug: hypertrombopa — In group A, they were treated with rhTPO and hypertrombopa, and were medicated until their PLT was ≥75×109/L. In group B, they were treated with rhTPO and hypertrombopa, and were medicated until their PLT was ≥75×109/L.

SUMMARY:
This study was an open-label, controlled, single-center, prospective phase II trial. In this prospective, real-world study, consecutive patients meeting eligibility criteria will be enrolled and allocated to: Group A (Grade Ⅱ CTIT, PLT:50-75*10^9/L) and Group B (Grade Ⅲ or higher CTIT，PLT:<50*10^9/L). Both groups received rhTPO and Hetrombopag treatment. A target sample size of 100 participants will be observed to characterize the clinical features and treatment patterns of cancer therapy-induced thrombocytopenia. Recombinant human thrombopoietin (rhTPO) and hetrombopag will be administered until a platelet count ≥ 75 × 10⁹/L is achieved. Beyond the protocol-specified dual therapy, basic management, including supportive care or concomitant medications-will remain at the investigator's discretion.

DETAILED DESCRIPTION:
This research will gather real-world data on an investigational drug in a prospective manner, aiming to monitor 100 patients to explore the characteristics and treatment approaches of thrombocytopenia associated with tumor therapy. In this prospective, real-world study, consecutive patients meeting eligibility criteria will be enrolled and allocated to: Group A (Grade Ⅱ CTIT, PLT:50-75*10^9/L) and Group B (Grade Ⅲ or higher CTIT，PLT:<50*10^9/L).

Patients with platelet counts between 50×10^9/L and 75×10^9/L will be randomly allocated to either Arm A or Arm B. In Arm A and Arm B, participants will receive standard care, which may include medications such as interleukin-11, leucogen, and yixuesheng. Meanwhile, individuals in Arm B will be administered recombinant human thrombopoietin (rhTPO) and eltrombopag until their platelet count reaches or exceeds 75×10^9/L.

This study will prospectively gather relevant patient information. Data collection will occur over two tumor treatment cycles and during the administration of thrombopoietin-promoting drugs for all participants. Specifically, the following data will be collected for each patient across two consecutive chemotherapy cycles (Cycle N and Cycle N+1):

* Patient baseline characteristics
* Dosage, frequency, and duration of administration for each study drug
* Details of concomitant medications related to the study drugs, including names, dosages, frequencies, and durations of administration
* Laboratory test results and imaging examination findings before, during, and after treatment with each study drug
* Records of any adverse events

The aim is to comprehensively document these aspects to ensure thorough analysis and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Understand the study procedures and voluntarily sign the informed consent form to voluntarily enroll in this study;
* Age ≥ 18 years old;
* Receive anti-tumor therapy (including chemotherapy, targeted therapy, immunotherapy, etc.) within 14 days prior to study entry;
* Anti-tumor therapy (see the subsequent 'Protocols for Reference' for details);
* Patients with two consecutive platelet counts <75×109/L more than 24 hours apart, with a screening period of 3 days.

Exclusion Criteria:

* Previous use of rhTPO or TPORA analogs;
* Prior grade 2 or higher CTIT;
* Patients undergoing clinical interventional studies;
* Patients with a history of hematologic malignancies, including leukemia, myeloma, myeloproliferative disorders, lymphoma, or myelodysplastic disorders;
* Patients with underlying liver disease (e.g., cirrhosis or chronic hepatitis) and no primary or metastatic cancer in the liver will be excluded if ALT/AST >3X ULN or total bile >3X ULN);
* Patients with the presence of primary or metastatic liver cancer will be excluded if ALT/AST >5X ULN or total bile >5X ULN;
* Patients with a history of symptomatic venous thrombotic events (e.g., DVT or pulmonary embolism) and symptomatic arterial thrombotic events (e.g., myocardial infarction, ischemic cerebral vascular accident, or transient ischemic attack) who are unable to tolerate anticoagulant therapy will be ineligible, and patients with D-dimer greater than 10,000 g/L will also be excluded;
* Serious concomitant medical conditions that may interfere with the conduct of the clinical trial, such as unstable angina, renal failure requiring hemodialysis, or active infection requiring intravenous antibiotics;
* Pregnant/nursing mothers and patients who do not wish to use contraception; Inability to understand the research nature of the study or failure to obtain informed consent;
* Other conditions that, in the judgment of the investigator, make inclusion in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumor therapy-related thrombocytopenia treated with thrombopoietic agents
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time for platelets to rise from nadir to 75 x 109/L | up to 4 weeks
  Time for platelets to rise from nadir to 75 x 109/L

SECONDARY OUTCOMES:
The time required for platelet count to rise to 100×10⁹/L, the proportion of patients with a delay of ≥7 days in the next cycle, bleeding, receiving platelet transfusion and treatment-related adverse reactions. | up to 4 weeks
  The time required for platelet count to rise to 100×10⁹/L, the proportion of patients with a delay of ≥7 days in the next cycle, bleeding, receiving platelet transfusion and treatment-related adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfei Fu, PhD, Principal Investigator — Director of Medical Oncology Department of Jinhua Municipal Central Hospital
Locations (1):
- Jinhua Central Hospital, Jinhua, Zhejiang, China